CLINICAL TRIAL: NCT04435366
Title: A Phase 3 Multicenter, Randomized, Double Masked, Sham- Controlled Clinical Trial to Assess the Safety and Efficacy of Intravitreal Administration of Zimura (Complement C5 Inhibitor) in Patients With Geographic Atrophy Secondary to Age-Related Macular Degeneration
Brief Title: A Phase 3 Safety and Efficacy Study of Intravitreal Administration of Zimura (Complement C5 Inhibitor)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IVERIC bio, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISEE2008
Record Dates: First submitted 2020-05-12; First posted 2020-06-17 (Actual); Results first posted 2023-12-28 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Geographic Atrophy; Macular Degeneration
Keywords: Geographic Atrophy (GA); Age-related Macular Degeneration; AMD; Complement C5 inhibitor; avacincaptad pegol; IZERVAY
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant, "Evaluating" Investigator, Reading Center Personnel, and Sponsor Personnel are masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Avacincaptad Pegol (Experimental): Participants received avacincaptad pegol (ACP) 2 milligram (mg)/eye via intravitreal (IVT) injections monthly through Month 11 (Year 1). At month 12, participants were re-randomized to receive ACP 2 mg/eye via IVT injections monthly from month12 through month 23 (Year 2).
  Interventions: Drug: Avacincaptad Pegol
- Sham (Sham Comparator): Participants received sham injections; through Month 11 (Year 1). At month 12, participants continued to receive monthly sham administration from month 12 through month 23 (Year 2).
  Interventions: Drug: Sham
- Avacincaptad pegol and Sham (Experimental): Participants who received ACP 2mg monthly through Month 11 (Year 1) were re-randomized at month 12, to receive ACP 2 mg/eye via IVT injections every other month at months 13, 15, 17, 19, 21, and 23 and sham injections at months 12, 14, 16,18, 20, and 22.
  Interventions: Drug: Avacincaptad Pegol

INTERVENTIONS:
Drug: Avacincaptad Pegol — Avacincaptad Pegol Intravitreal Injection
  Other Names: Zimura (previous name); IZERVAY
  Arms: Avacincaptad Pegol; Avacincaptad pegol and Sham
Drug: Sham — Sham Administration (includes placement of the blunt opening of an empty, needleless syringe barrel on the conjunctiva in the inferotemporal quadrant of the eyeball to simulate the pressure of an injection)
  Arms: Sham

SUMMARY:
The objectives of this study was to evaluate the safety and efficacy of avacincaptad pegol intravitreal administration in participants with geographic atrophy secondary to age-related macular degeneration (AMD)

DETAILED DESCRIPTION:
Participants were randomized in a 1:1 ratio to the following monthly treatment groups:

* Avacincaptad pegol 2 mg
* Sham

At Month 12, the participants in the avacincaptad pegol 2mg treatment group were re-randomized to receive the study drug either on a monthly basis or on an every other month basis

The participants initially randomized to sham treatment continued with monthly sham administration through Month 23

All participants had a final follow up visit at Month 24

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender aged ≥ 50 years
* Diagnosis of Non-foveal GA secondary to dry AMD

Exclusion Criteria:

* Any prior treatment for AMD (dry or wet) or any prior intravitreal treatment for any indication in either eye, except oral supplements of vitamins and minerals
* Any intraocular surgery or thermal laser within 3 months of trial entry.
* Any prior thermal laser in the macular region, regardless of indication
* Any ocular or periocular infection (including blepharitis), or ocular surface inflammation in the past 12 weeks.
* Previous therapeutic radiation in the region of the study eye
* Any sign of diabetic retinopathy in either eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2023-08-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (205):
- United States (96):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Retinal Diagnostic Center, Campbell, California
  - Eye Medical Center of Fresno, Fresno, California
  - Retina Consultants of Orange County, Fullerton, California
  - University of California, San Diego, La Jolla, California
  - Jules Stein Eye Institute/David Geffen School of Medicine, Los Angeles, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - California Retina Consultants, Oxnard, California
  - Southern California Desert Retina Consultants, Palm Desert, California
  - Doheny Eye Center, UCLA, Pasadena, California
  - Retina Consultants of Southern California, Redlands, California
  - Retinal Consultants Medical Group, Inc., Sacramento, California
  - Orange County Retinal Medical Group, Santa Ana, California
  - University of Colorado, Aurora, Colorado
  - Retina Consultants of Southern Colorado, P.C., Colorado Springs, Colorado
  - Colorado Retina Associates, Lakewood, Colorado
  - Connecticut Eye Consultants, P.C., Danbury, Connecticut
  - Retina Group of New England, PC, Waterford, Connecticut
  - Florida Eye Clinic, Altamonte Springs, Florida
  - Rand Eye Institute, Deerfield Beach, Florida
  - Retina Group of Florida, Fort Lauderdale, Florida
  - Retina Health Center, Fort Myers, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - VitreoRetinal Associates, P.A., Gainesville, Florida
  - Florida Eye Associates, Melbourne, Florida
  - University of Miami-Bascom Palmer Eye Institute, Miami, Florida
  - Retina Care Specialists, Palm Beach Gardens, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Retina Associates of Sarasota, Sarasota, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - East Florida Eye Institute, Stuart, Florida
  - Southern Vitreoretinal Associates, PL, Tallahassee, Florida
  - Center for Retina and Macula Disease, Winter Haven, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina, P.C., Marietta, Georgia
  - Retina Consultants of Hawaii, Inc, ‘Aiea, Hawaii
  - University Retina and Macula Associates, PC, Lemont, Illinois
  - Illinois Eye Center, Peoria, Illinois
  - Midwest Eye Institute, Indianapolis, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Retina Associates, LLC, Lenexa, Kansas
  - Vitreo Retinal Consultants & Surgeons, Wichita, Kansas
  - Ochsner Medical Center, New Orleans, Louisiana
  - The Retina Care Center, Baltimore, Maryland
  - The Retina Group of Washington, Chevy Chase, Maryland
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Retina Research Institute at New England Retinal Consultants, Springfield, Massachusetts
  - UMASS Memorial Eye Center, Worcester, Massachusetts
  - Vitreoretinal Associates, PC, Worcester, Massachusetts
  - Associated Retinal Consultants, P.C., Royal Oak, Michigan
  - Retina Center, Minneapolis, Minnesota
  - St. Louis University, St Louis, Missouri
  - Retina Consultants of Nevada, Henderson, Nevada
  - Sierra Eye Associates, Reno, Nevada
  - Retina Center of New Jersey, LLC, Bloomfield, New Jersey
  - Long Island Vitreoretinal Consultant, Great Neck, New York
  - Retina Vitreous Surgeons of Central New York, PC, Liverpool, New York
  - Vitreous Retina Macula Consultants of New York (VRMNY), New York, New York
  - OCLI, Oceanside, New York
  - Retina Associates of Western NY, PC, Rochester, New York
  - Ophthalmic Consultants of the Capital Region, Troy, New York
  - Western Carolina Retinal Associates, Asheville, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Retina and Vitreous Center of Southern Oregon, Ashland, Oregon
  - Retina Northwest, PC, Portland, Oregon
  - EyeHealth Northwest, Portland, Oregon
  - Casey Eye Institute, Portland, Oregon
  - Scheie Eye Institute, University of Pennsylvania, Philadelphia, Pennsylvania
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Associates in Ophthalmology, Ltd, West Mifflin, Pennsylvania
  - Retina Research of Beaufort, LLC, Beaufort, South Carolina
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Carolina Macula and Retina, Mt. Pleasant, South Carolina
  - Palmetto Retina Center, West Columbia, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Southeastern Retina Associates, PC, Johnson City, Tennessee
  - Southeastern Retina Associates, PC, Knoxville, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Southwest Retina Specialists, Amarillo, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Foundation of the Southwest, Dallas, Texas
  - Retina and Vitreous of Texas, PLLC, Houston, Texas
  - Valley Retina Institute, McAllen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Center of Texas, Southlake, Texas
  - Retinal Consultants of Houston, The Woodlands, Texas
  - Strategic Clinical Research Group, Willow Park, Texas
  - Retinal Associates of Utah, Salt Lake City, Utah
  - Rocky Mountain Retina Consultants, Salt Lake City, Utah
  - University of Utah, John A. Moran Eye Center, Salt Lake City, Utah
  - Wagner Macular & Retina Center, Norfolk, Virginia
  - Retina Institute of Virginia, Richmond, Virginia
  - Vistar Eye Center, Roanoke, Virginia
  - Pacific Northwest Retina, Bellevue, Washington
  - Retina Center NW, PLLC, Silverdale, Washington
- Argentina (9):
  - Centro Oftalmológico Dr. Charles SA, Buenos Aires, Buenos Aires F.D.
  - Buenos Aires Macula S.A., Buenos Aires, Buenos Aires F.D.
  - Centro Médico Grupo Laser Visión, Rosario, Santa Fe Province
  - Centro de Diagnóstico y Cirugía Ocular "Oftalmólogos Especialistas", Rosario, Santa Fe Province
  - Instituto Oftalmológico de Buenos Aires, Buenos Aires
  - Centro Privado de Ojos Romagosa S.A., Córdoba
  - Instituto Oftalmológico de Córdoba, Córdoba
  - Centro Privado de Oftalmologia - OFTAR Mendoza SRL, Mendoza
  - Centro Medico Micro Diagnostico y Microcirugla Ocular, Rosario
- Australia (3):
  - Sydney Eye Hospital, Sydney, New South Wales
  - Sydney Retina Clinic and Day Surgery, Sydney, New South Wales
  - Royal Victorian Eye & Ear Hospital, East Melbourne
- Austria (4):
  - Medizinische Universitaet Graz - Augenklinik, Graz
  - Medizinische Universitaet Innsbruck - Universitaetsklinik fuer Augenheilkunde und Optometrie, Innsbruck
  - Medical University of Vienna, Vienna
  - Hanush Hospital, Vienna
- CHU Brugmann, Brussels, Belgium
- Brazil (3):
  - Centro de Ensino e Pesquisa do Instituto da Visao (CEPIV), Belo Horizonte
  - IPEPO - Instituto da visão, São Paulo
  - Hospital Sao Paulo - UNIFESP, Vila Clementino
- Canada (7):
  - Calgary Retina Consultants, Calgary, Alberta
  - UBC/VGH Eye Care Center, Vancouver, British Columbia
  - St.Joseph's Health Care London, London, Ontario
  - Canadian Centre for Advanced Eye Therapeutics Inc., Mississauga, Ontario
  - University of Ottawa Eye Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - Retina Centre of Ottawa, Ottawa
- Colombia (2):
  - Clinica De Oftalmologia Sandiego, Medellín, Antioquia
  - Fundacion OJlalmologica Nacional - FUNDONAL, Bogotá
- Clinical hospital Center Osijek, Osijek, Croatia
- Axon Clinical s.r.o., Prague, Smichov, Czechia
- Estonia (2):
  - Dr Kai Noor Silmakabinet, Tallinn
  - Tartu University Hospital, Tartu
- France (13):
  - CHU de Bordeaux - Hopital Pellegrin, Bordeaux
  - Hopital Intercommunal, Créteil
  - CHU Bocage, Dijon
  - Centre Pole Vision Val d'Ouest, Écully
  - Centre d'ophtalmologie Rabelais, Lyon
  - Hopital de la Croix Rousse, Lyon
  - Centre Paradis Monticelli, Marseille
  - CHU de Nantes, Nantes
  - Centre d'exploration ophtalmologique de l'Odeon, Paris
  - Hôpital Lariboisière, Paris
  - Centre Ophtalmologique d'Imagerie et de Laser, Paris
  - Fondation Alolphe de Rotschild, Paris
  - Centre St Exupery, Saint-Cyr-sur-Loire
- Germany (14):
  - RWTH Aachen University, Aachen
  - University of Bonn, Bonn
  - Augenklinik University Hospital Cologne, Cologne
  - University of Göttingen, Göttingen
  - Universitätsklinikum Hamburg Eppendorf Klinik und Poliklinik für Augenheilkunde Studienzentrum, Hamburg
  - University Eye Hospital, MHH, Hanover
  - University clinic Leipzig AÖR, Leipzig
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Ludwig-Maximilians-University Munich, Munich
  - Clinic Rechts der Isar, Munich
  - Augenzentrum am St. Franziskus-Hospital, Münster
  - Universitätsklinikum Münster, Münster
  - Universitäts-Augenklinik, Tübingen
- Hungary (8):
  - Hungarian Military Hospital Center, Budapest
  - Bajcsy Zsilinszky Kórház - Szemészet, Budapest
  - Budapest Retina Associates, Budapest
  - Semmelweis University, Dept of Ophthalmology, Budapest
  - Debrecen University Clinical Center, Dept of Ophthalmology, Debrecen
  - Szabolcs-Szatmar-Bereg County Hospital and University Teaching Hospital, Nyíregyháza
  - Ganglion Medical Center, Pécs
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
- Israel (9):
  - Barzilai Medical Center, Ashkelon
  - Shamir Medical Center, Be’er Ya‘aqov
  - Rambam Medical Centre, Haifa
  - Carmel Medical Center, Haifa
  - Edith Wolfson Medical Center, Holon
  - Hadassah University Hospital, Jerusalem
  - Department of Ophthalmology, Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Sourasky Medical Center, Tel Aviv
- Italy (14):
  - Ospedali Riuniti di Ancona, Ancona
  - A.O.U. Policlinico Sant'Orsola-Malpighi, Bologna
  - Ospedale Clinicizzato Universita di Chieti "Ss Annunziata", Chieti
  - Nuovo Arcispedale Sant' Anna (A.O.U. di Ferrara), Ferrara
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale Maggiore Policlinico Milano, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Ospedale Luigi Sacco, Milan
  - AOU Universita degli Studi della Campania Luigi Vanvitelli UOC Oculistica, Naples
  - Azienda Ospedaliera di Padova Unità Operativa Complessa di Clinica Oculistica, Padua
  - University of Pisa, Pisa
  - Fondazione PTV, Roma
  - Fondazione GB Bietti IRCCS, Roma
  - Azienda Sanitaria Universitaria Integrata, Udine
- Pauls Stradinis Clinical University Hospital, Riga, Latvia
- Poland (4):
  - Klinika Okulistyczna OFT ALMIKA Sp. z o. o., Bydgoszcz
  - Medical Center Julianów, Lodz
  - Caminomed, Tarnowskie Góry
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego, Wroclaw
- Spain (12):
  - Clinica de Oftalmologia Barraquer, Barcelona
  - Institut Catala de Retina, Barcelona
  - Institut de la Macula, Barcelona
  - VOR - Hospital General de Catalunya, Barcelona
  - Instituto Clinico Quirurgico de Oftalmologia, Bilbao
  - Hospital La Arruzafa, Córdoba
  - H.U. Puerta de Hierro-Majadahonda, Majadahonda
  - Clinica Universidad de Navarra, Pamplona
  - Instituto Oftalmologico Gomez-Ulla, Santiago de Compostela
  - IMED Servicio Oftalmología, Valencia
  - Rio Hortega University Hospital, Valladolid
  - Hospital Clínico Universitario "Lozano Blesa", Zaragoza
- Hull University Teaching Hospitals NHS Trust, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Khanani AM, Danzig CJ, Heier JS, Jaffe GJ, Kaiser PK, Lally DR, Patel SS, Vajzovic L, Weng CY, Patel H, Clark J, Desai D, Luo D, Henry E, Holz FG; GATHER2 trial investigators. Avacincaptad pegol for geographic atrophy secondary to age-related macular degeneration: 2-year efficacy and safety results from the GATHER2 phase 3 trial. Ophthalmology. 2025 Dec 15:S0161-6420(25)00790-0. doi: 10.1016/j.ophtha.2025.12.011. Online ahead of print. PMID 41407269
- [Derived] Khanani AM, Patel SS, Staurenghi G, Tadayoni R, Danzig CJ, Eichenbaum DA, Hsu J, Wykoff CC, Heier JS, Lally DR, Mones J, Nielsen JS, Sheth VS, Kaiser PK, Clark J, Zhu L, Patel H, Tang J, Desai D, Jaffe GJ; GATHER2 trial investigators. Efficacy and safety of avacincaptad pegol in patients with geographic atrophy (GATHER2): 12-month results from a randomised, double-masked, phase 3 trial. Lancet. 2023 Oct 21;402(10411):1449-1458. doi: 10.1016/S0140-6736(23)01583-0. Epub 2023 Sep 8. PMID 37696275
- [Derived] Tzoumas N, Riding G, Williams MA, Steel DH. Complement inhibitors for age-related macular degeneration. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD009300. doi: 10.1002/14651858.CD009300.pub3. PMID 37314061
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website. — https://www.clinicaltrials.astellas.com/study/ISEE2008/
- See also: Link to plain language summary of the study on the Trial Results Summaries website. — https://www.trialsummaries.com/Study/StudyDetails?id=26044&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants ≥ 50 years of age diagnosed with geographic atrophy (GA) that was at least partly within 1.5 mm radius from the foveal center were enrolled in the study.
Pre-assignment Details: Participants who met all inclusion criteria and none of the exclusion criteria were enrolled in the study.
Groups:
- Avacincaptad Pegol: Participants received ACP 2 mg/eye via IVT injections monthly through Month 11 (Year 1). At month 12, participants were re-randomized to receive ACP 2 mg/eye via IVT injections monthly from month12 through month 23 (Year 2). Participants were followed up until month 24.
- Avacincaptad Pegol and Sham: Participants received ACP 2 mg/eye via IVT injections monthly through Month 11 (Year 1). At month 12, participants were re-randomized to receive ACP 2 mg/eye via IVT every other month (EOM) at months 13, 15, 17, 19, 21, and 23 and sham injections at months 12, 14, 16,18, 20, and 22 (Year 2). Participants were followed up until month 24.
- Sham: Participants received sham injections; through Month 11 (Year 1). At month 12, participants continued to receive monthly sham injection from month 12 through month 23 (Year 2). Participants were followed up until month 24.
Period: Year 1 (12 Months)
Arm/Group | Avacincaptad Pegol | Avacincaptad Pegol and Sham | Sham
Started | 225 | 0 | 223
Treated | 225 | 0 | 222
Completed | 200 | 0 | 205
Not Completed | 25 | 0 | 18
Not completed — Adverse Event | 3 | 0 | 2
Not completed — Death | 2 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 1
Not completed — Withdrawal by Subject | 17 | 0 | 13
Not completed — Patient non-compliance | 1 | 0 | 0
Not completed — Not treated | 0 | 0 | 1
Period: Year 2 (12 Months)
Arm/Group | Avacincaptad Pegol | Avacincaptad Pegol and Sham | Sham
Started | 96 | 93 | 203
Completed | 89 | 83 | 184
Not Completed | 7 | 10 | 19
Not completed — Death | 1 | 4 | 6
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Withdrawal by Subject | 4 | 3 | 7
Not completed — Adverse Event | 2 | 1 | 6

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set consisted of all randomized participants who received at least 1 dose of study drug.
Groups:
- Avacincaptad Pegol: Participants received ACP 2 mg/eye via IVT injections monthly through Month 11 (Year 1). At month 12, participants were re-randomized to receive ACP 2 mg/eye via IVT injections monthly or ACP 2 mg/eye via IVT injections EOM at months 13, 15, 17, 19, 21, and 23 and sham injections at months 12, 14, 16,18, 20, and 22 (Year 2). Participants were followed up until month 24.
- Total: Total of all reporting groups
Arm/Group | Avacincaptad Pegol | Sham | Total
Number analyzed (Participants) | 225 | 222 | 447
Age, Continuous [Mean (Standard Deviation); unit: Years] | 76.3 (8.6) | 76.7 (8.8) | 76.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 156 | 310
  Male | 71 | 66 | 137
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 23 | 50
  Not Hispanic or Latino | 168 | 178 | 346
  Unknown or Not Reported | 30 | 21 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 182 | 186 | 368
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 41 | 34 | 75

OUTCOME MEASURES:

1. Primary Outcome: The Mean Rate of Growth (Slope) Estimated Based on GA Area Measured by Autofluorescence (FAF) at 3 Time Points: Baseline, Month 6, and Month 12
Description: GA was associated with age-related macular degeneration (AMD) and caused bilateral, progressive, and irreversible loss of retinal tissue (photoreceptors, retinal pigment epithelium, and choriocapillaris) leading to a permanent loss of visual function and blindness. The least squares mean used to determine mean rate of change in GA growth (slope) was measured by FAF. LS mean & SE were based on square-root transformation.
Time Frame: Baseline to month 12
Population: ITT analysis set
Measure: Least Squares Mean (Standard Error); unit: millimeters (mm)/year
Arm/Group | Avacincaptad Pegol | Sham
Number analyzed (Participants) | 225 | 222
millimeters (mm)/year | 0.336 (0.032) | 0.392 (0.033)
Statistical Analysis 1: Comparison: Avacincaptad Pegol vs Sham; Difference in least squares mean between groups calculated as (sham) minus (avacincaptad pegol). Mixed Model for repeated measures (MMRM) was used to compare the treatment groups; Test type: Superiority; p = 0.0064, MMRM — Nominal p-value was used for the comparison between avacincaptad pegol versus sham; Least Squares Mean Difference = 0.056, 95% CI 2-sided [0.016 to 0.096], Standard Error of Mean 0.020

2. Primary Outcome: The Mean Rate of Growth (Slope) Estimated Based on GA Area Measured by FAF at 5 Timepoints: Baseline, Month 6, Month 12, Month 18, and Month 24
Description: GA was associated with AMD and caused bilateral, progressive, and irreversible loss of retinal tissue (photoreceptors, retinal pigment epithelium, and choriocapillaris) leading to a permanent loss of visual function and blindness. The least square mean rate of GA growth (slope) was measured by FAF. LS mean & SE were based on untransformed data.
Time Frame: Baseline to month 24
Population: Re-rand analysis set-The subset of the ITT analysis set who were re-randomized at Month 12 and who were on sham and completed the Month 12 visit.
Measure: Least Squares Mean (Standard Error); unit: mm^2/year
Arm/Group | Avacincaptad Pegol | Avacincaptad Pegol and Sham | Sham
Number analyzed (Participants) | 96 | 93 | 222
mm^2/year | 2.23 (0.124) | 2.10 (0.126) | 2.59 (0.085)
Statistical Analysis 1: Comparison: Avacincaptad Pegol vs Sham; Difference in least squares mean between groups calculated as (sham) minus (avacincaptad pegol); Test type: Superiority; p = 0.0165, MMRM — Nominal p-value was used for the comparison between avacincaptad pegol versus sham; Least Squares Mean Difference = 0.362, 95% CI 2-sided [0.066 to 0.657], Standard Error of Mean 0.150
Statistical Analysis 2: Comparison: Avacincaptad Pegol and Sham vs Sham; Difference in least squares mean between groups calculated as (sham) minus (avacincaptad pegol and sham); Test type: Superiority; p = 0.0015, MMRM — Nominal p-value was used for the comparison between avacincaptad pegol and sham versus sham; Least Squares Mean Difference = 0.488, 95% CI 2-sided [0.189 to 0.788], Standard Error of Mean 0.152

3. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) Using Early Treatment Diabetic Retinopathy Study (ETDRS) Letters at 24 Months
Description: BCVA was assessed using ETDRS visual acuity testing charts. The ETDRS Visual Acuity Score (VAS) is defined as the number of letters read on the ETDRS chart. Minimum and maximum possible scores are 0-100. A higher score represented better visual functioning. A positive change from baseline indicates an improvement and a negative change from baseline indicates a worsening.
Time Frame: Baseline and month 24
Population: ITT analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Avacincaptad Pegol | Sham
Number analyzed (Participants) | 225 | 222
score on a scale | -7.31 (1.07) | -6.48 (1.05)
Statistical Analysis 1: Comparison: Avacincaptad Pegol vs Sham; Difference in least squares mean between groups calculated as (sham) minus (avacincaptad pegol); Test type: Superiority; p = 0.58, MMRM — Nominal p-value was used for the comparison between avacincaptad pegol versus sham; Least Squares Mean Difference = -0.83, 95% CI 2-sided [-3.79 to 2.12], Standard Error of Mean 1.50

4. Secondary Outcome: Change From Baseline in Low Luminance (LL) BCVA Using ETDRS Letters at 24 Months
Description: BCVA was assessed using ETDRS visual acuity testing charts. The ETDRS VAS is defined as the number of letters read on the ETDRS chart. Minimum and maximum possible scores are 0-100. A higher score represented better visual functioning. A positive change from baseline indicates an improvement and a negative change from baseline indicates a worsening. LL BCVA was measured by placing a 2.0 log unit neutral density filter over the best correction for that eye and having the participant read the normally illuminated ETDRS chart.
Time Frame: Baseline and month 24
Population: ITT analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Sham: Participants received sham injections; through Month 11 (Year 1). At month 12, participants continued to receive monthly sham injection from month 12 through month 23 (Year 2). ). Participants were followed up until month 24.
Arm/Group | Avacincaptad Pegol | Sham
Number analyzed (Participants) | 225 | 222
score on a scale | -10.58 (1.20) | -9.1 (1.18)
Statistical Analysis 1: Comparison: Avacincaptad Pegol vs Sham; Difference in least squares mean between groups calculated as (sham) minus (avacincaptad pegol); Test type: Superiority; p = 0.38, MMRM — Nominal p-value was used for the comparison between avacincaptad pegol versus sham; Least Squares Mean Difference = -1.49, 95% CI 2-sided [-4.79 to 1.81], Standard Error of Mean 1.68

5. Secondary Outcome: Change From Baseline in Visual Function Questionnaire (VFQ-25) Composite Scores at 6, 12 and 18 Months
Description: The National Eye Institute Visual Function Questionnaire-25 (VFQ-25) measured the influence of visual disability and visual symptoms on general health domains. The VFQ-25 consisted of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question. A higher score represented better visual functioning. Each item was then converted to a 0 to 100 scale so that the lowest and highest possible scores were set at 0 and 100 points, respectively. Each subscale score had a range of 0 to 100 inclusive and were calculated from the re-scaled raw data. A composite score was derived based on the average of the 11 vision-related subscales.
Time Frame: Baseline, months 6, 12, and 18
Population: ITT analysis set with available data was analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Avacincaptad Pegol | Sham
Number analyzed (Participants) | 206 | 215
score on a scale
  Change at 6 months | -1.2 (10.56) | -1.6 (9.98)
  Change at 12 months: number analyzed (Participants) | 196 | 199
  Change at 12 months | -3.4 (11.05) | -3.6 (11.01)
  Change at 18 months: number analyzed (Participants) | 173 | 187
  Change at 18 months | -5.4 (12.80) | -4.7 (11.53)

6. Secondary Outcome: Change From Baseline in Visual Function Questionnaire (VFQ-25) Composite Scores at 24 Months
Description: as for outcome 5
Time Frame: Baseline and month 24
Population: ITT analysis
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Avacincaptad Pegol | Sham
Number analyzed (Participants) | 225 | 222
score on a scale | -7.735 (0.950) | -7.023 (0.931)
Statistical Analysis 1: Comparison: Avacincaptad Pegol vs Sham; Test type: Superiority; p = 0.5929, MMRM; Least square mean difference = -0.712, 95% CI 2-sided [-3.326 to 1.903], Standard Error of Mean 1.330

7. Secondary Outcome: Number of Participants With Categorical One-level Loss in VFQ-25 Subscale
Description: The National Eye Institute VFQ-25 measured the influence of visual disability and visual symptoms on general health domains. The VFQ-25 consisted of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question. A higher score represented better visual functioning. Each item was then converted to a 0 to 100 scale so that the lowest and highest possible scores were set at 0 and 100 points, respectively.Categorical one-level loss in each item was defined as decline of one or more levels at Month 24 on the original scale from Baseline (equivalently 20 points for general vision and 25 points for other vision items in a 0 to 100 scale).
Time Frame: Baseline up to month 24
Population: ITT analysis set with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Avacincaptad Pegol | Sham
Number analyzed (Participants) | 175 | 182
participants
  Color Vision | 45 | 35
  Distance Vision | 56 | 43
  Near Vision | 61 | 49
  Peripheral Vision | 58 | 65
  General Vision | 58 | 58
  Dependency | 55 | 55
  Driving | 27 | 26
  General Health | 45 | 67
  Mental Health | 35 | 42
  Ocular Pain | 27 | 20
  Role Difficulties | 60 | 59
  Social Function | 52 | 52

8. Secondary Outcome: Time to Persistent Vision Loss
Description: Vision loss event was defined as a loss of ≥ 15 letters (equivalent to a loss of 3 lines on the ETDRS chart) in BCVA from Baseline measured at any two or more consecutive visits up to Month 24. These parameters were chosen as a 3-line BCVA loss (equivalent to doubling of visual angle) is widely recognized as a significant deterioration in vision and a minimum of two consecutive visits was representative of persistent disease progression. BCVA was assessed using ETDRS visual acuity testing charts. The ETDRS VAS was defined as the number of letters read on the ETDRS chart. Min and max possible scores are 0-100. A higher score represents better visual functioning. Kaplan-Meier method was used for analysis. Participants with an event were reported and not the median time to event.
Time Frame: Baseline up to month 24
Population: ITT analysis set
Measure: Median (Full Range); unit: months
Arm/Group | Avacincaptad Pegol | Sham
Number analyzed (Participants) | 225 | 222
months | 17.02 [2.8 to 23.0] | 13.93 [1.3 to 23.2]
Statistical Analysis 1: Comparison: Avacincaptad Pegol vs Sham; Test type: Superiority; p = 0.6424, Log Rank; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.57 to 1.42]

ADVERSE EVENTS:
Time Frame: All-cause mortality (ACM): From randomization up to 24 months Serious Adverse events (SAEs) and non-SAEs: From first dose up to 24 months
Description: Participants in "ACP only" & "ACP and Sham" groups were treated with ACP for up to 2 years, hence safety of ACP is more accurately represented by the randomized ACP group.
  ACM: All randomized participants. Serious & non-SAEs: Those who received at least 1 dose of treatment. Those who received injection of ACP were analyzed in ACP group according to actual injections. One participant randomized to sham didn't receive treatment & was included in denominator for ACM only and not for other outcomes.
Groups:
- Avacincaptad Pegol Only (up to 12 Months): Participants received ACP 2 mg/eye via IVT injections monthly through Month 11 (Year 1).
- Avacincaptad Pegol Only (12 to 24 Months): Participants were re-randomized at month 12 to receive ACP 2 mg/eye via IVT injections monthly from month 12 through month 23 (Year 2). Participants were followed up until month 24.
- Avacincaptad Pegol and Sham Only (12 to 24 Months): Participants were re-randomized at month 12, to receive ACP 2 mg/eye via IVT injections every other month at months 13, 15, 17, 19, 21, and 23 and sham injections at months 12, 14, 16,18, 20, and 22 (Year 2). Participants were followed up until month 24.
- Sham Only (up to 12 Months): Participants received sham injections through Month 11 (Year 1).
- Sham Only (12 to 24 Months): Participants continued to receive monthly sham injection from month 12 through month 23 (Year 2). Participants were followed up until month 24.
Arm/Group | Avacincaptad Pegol Only (up to 12 Months) | Avacincaptad Pegol Only (12 to 24 Months) | Avacincaptad Pegol and Sham Only (12 to 24 Months) | Sham Only (up to 12 Months) | Sham Only (12 to 24 Months)
All-Cause Mortality (participants affected / at risk) | 4/225 | 1/96 | 4/93 | 1/222 | 7/203
Serious Adverse Events (participants affected / at risk) | 31/225 | 18/96 | 16/93 | 36/222 | 25/203
Other Adverse Events (participants affected / at risk) | 100/225 | 51/96 | 41/93 | 83/222 | 77/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avacincaptad Pegol Only (up to 12 Months) (N=225) | Avacincaptad Pegol Only (12 to 24 Months) (N=96) | Avacincaptad Pegol and Sham Only (12 to 24 Months) (N=93) | Sham Only (up to 12 Months) (N=222) | Sham Only (12 to 24 Months) (N=203)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery insufficiency (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mobile caecum syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Choroidal neovascularisation (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual acuity reduced transiently (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis intestinal perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endophthalmitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Listeria sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-small cell lung cancer stage IIIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinonasal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Neuromyelitis optica spectrum disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device lead damage (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neurogenic shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avacincaptad Pegol Only (up to 12 Months) (N=225) | Avacincaptad Pegol Only (12 to 24 Months) (N=96) | Avacincaptad Pegol and Sham Only (12 to 24 Months) (N=93) | Sham Only (up to 12 Months) (N=222) | Sham Only (12 to 24 Months) (N=203)
Cataract (Eye disorders) | 6 (8) | 7 (8) | 4 (5) | 9 (13) | 10 (13)
Choroidal neovascularisation (Eye disorders) | 21 (21) | 11 (13) | 8 (8) | 11 (13) | 19 (21)
Conjunctival haemorrhage (Eye disorders) | 31 (55) | 14 (22) | 9 (16) | 18 (32) | 5 (8)
Conjunctival hyperaemia (Eye disorders) | 12 (34) | 1 (1) | 1 (1) | 13 (38) | 5 (6)
Punctate keratitis (Eye disorders) | 14 (25) | 5 (8) | 5 (6) | 15 (32) | 5 (14)
Retinal haemorrhage (Eye disorders) | 8 (9) | 2 (2) | 5 (6) | 5 (5) | 2 (3)
COVID-19 (Infections and infestations) | 7 (7) | 11 (11) | 14 (14) | 7 (7) | 26 (27)
Nasopharyngitis (Infections and infestations) | 4 (4) | 4 (6) | 6 (6) | 6 (8) | 3 (3)
Urinary tract infection (Infections and infestations) | 14 (17) | 3 (3) | 2 (2) | 13 (13) | 18 (22)
Fall (Injury, poisoning and procedural complications) | 14 (15) | 9 (9) | 8 (8) | 17 (18) | 12 (17)
Intraocular pressure increased (Investigations) | 22 (43) | 9 (18) | 5 (7) | 4 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No individual site or investigator may publish or present any results from the trial until a joint, multi-center publication of the trial results is made by Sponsor in conjunction with various participating investigators and appropriate sites contributing data and comments. Subsequently, individual investigators may request to publish or present results from the trial; however approval will be at the sole discretion of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/66/NCT04435366/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT04435366/SAP_002.pdf